CLINICAL TRIAL: NCT06956053
Title: Personalized Optimization of Antibiotic Therapy in Pulmonary Sepsis Critically Ill Patients Through Application of Rapid Microbiological Diagnostic Technologies and Pharmacokinetic/Pharmacodynamic Modelling
Acronym: IDAST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP180673
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Sepsis
Keywords: Pulmonary sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid ID/AST method (Experimental)
  Interventions: Diagnostic Test: Rapid ID/AST method
- Conventional microbiological methods (Active Comparator)
  Interventions: Diagnostic Test: Conventional biological methods

INTERVENTIONS:
Diagnostic Test: Rapid ID/AST method — 1. BioFire® Film Array® Blood Culture Identification 2 BCID2 panel, bioMérieux/BioFire Diagnostics, CE marked (FDA cleared)
  2. BioFire® FilmArray® Pneumonia Panels, CE marked (FDA cleared)
  3. SPECIFIC REVEAL® Rapid Antimicrobial Susceptibility test (AST) System, bioMérieux/Specific Diagnostics, CE-IVD and -IVDR marked
  Arms: Rapid ID/AST method
Diagnostic Test: Conventional biological methods — Usual care
  Arms: Conventional microbiological methods

SUMMARY:
Severe community-acquired and nosocomial pneumonia are associated with substantial morbidity and mortality. Early and appropriate antimicrobial therapy (AAT) is consistently the most effective intervention for reducing mortality. Cure is most likely when pharmacokinetic (PK) / pharmacodynamics (PD) targets associated with maximum antibiotic (ABX) activity are achieved. However, the process of optimizing antibiotic therapy for critically ill patients remains a complicated challenge.

A key issue is pathogen identification (ID) with subsequent antibiotic susceptibility testing (AST) results which allow for selection of AAT. Standard laboratory procedures typically require 2-3 days to provide ID and AST results. Optimal ABX dosing/dosing intervals depend in large part on PK properties in individual patients, and antibacterial effects on the infecting bacteria (PD). Alterations in the primary PK parameters, namely volume of distribution (Vd) and clearance (CL), are commonly observed, and are the most influential parameters in determining ABX dosing and exposure. ABX dosing/dosing intervals that do not account for these features are likely to lead to suboptimal ABX exposure and therapeutic failures. Because of 48-72-hours delays in ID/AST, initial treatment is frequently inappropriate in coverage, unnecessarily broad in spectrum, and/or suboptimal in dosing.

Methods for rapid bacterial growth, ID, AST and minimum inhibitory concentration (MIC) identification were developed and are capable of quantitative ID in 1-2 hours and major AST in 6-8 hours using clinical specimens. Rapid ID of the infecting pathogen and its individual AST could significantly impact the early selection of AAT and, combined with therapeutic drug monitoring data, could be used to calculate optimized dosing regimens that are personalized for the patient in order to achieve appropriate PK/PD targets.

Hypothesis: Application of these rapid ID/AST systems, together with prospective PK/PD monitoring of antibiotic plasma concentrations, will significantly shorten time from "sample to answer" for pathogen ID/AST, enhance personalized prescribing of antibiotics, optimize the time to targeted effective and AAT, and result in decreased treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in ICU
* 18 years of age or older
* With a pulmonary sepsis defined a s documented or suspected acute pulmonary infection (nosocomial and community-acquired pneumonia) and a SOFA score >2.
* Written Informed consent from the patient whenever possible or written ascent from next of kin whenever present at inclusion. When a patient would not be capable of consenting prior to randomization, his/her deferred consent will be gotten.

Exclusion Criteria:

* COVID-19 patients
* Severe anaphylactic beta-lactam allergy
* First measurements of prescribed antibiotic concentration (TDM) not possible within 24 hr after randomization
* Pregnancy or lactation
* Any decision of limitation of care
* Pre-existing medical condition with a life expectancy of less than 3 months
* Absence of affiliation to social security
* Patient under guardianship, curatorship and deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Rate of treatment failure | Up to 10 days after inclusion
  It includes treatment failure that occurred early (≤72 hours) or late (>72 hours), or at both times.

SECONDARY OUTCOMES:
Time to availability of pathogen | Up to 180 days
  ID/AST, MICs and conventional results
Time to achieve targeted optimized therapy | Up to 180 days
  It includes both pathogen-appropriate drug selection and appropriate dosing with plasma ABX concentration achieving PK/PD targets.
Time to antibiotic switches | Up to 180 days
Number of started, stopped, added or adjusted (escalation or de-escalation) antibiotics | Up to 180 days
Time to Aantibiotic dose adjustments to achieve PK/PD targets | Up to 180 days
All-Cause mortality | Up to 180 days
  At ICU
All-Cause mortality | Up to 180 days
  At hospital discharge
All Cause Mortality | At day 90
All Cause Mortality | At day 180
SOFA score assessment | Up to 28 days
  Evolution of organ failures by daily SOFA score assessment
Organ-failure free days (SOFA<6) | Up to day 28
Proportion of patients requiring invasive mechanical ventilation | At day 7
  Duration of invasive mechanical ventilation
Proportion of patients requiring invasive mechanical ventilation | At day 14
  Duration of invasive mechanical ventilation
Proportion of patients requiring invasive mechanical ventilation | At day 28
  Duration of invasive mechanical ventilation
Proportion of patients requiring invasive mechanical ventilation | At day 90
  Duration of invasive mechanical ventilation
Ventilator free days | At day 28
Vasopressor free days | At day 28
Vasopressor free days | At day 90
ICU length of stay | up to day 180
Hospital length of stay | up to day 180
Number of serious adverse events | up to day 180
  As per MEDDRA classification